CLINICAL TRIAL: NCT06679738
Title: Genetic Variants Associated With the Risk of Gall Stones and Cirrhosis.
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-67
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Liver Cirrhosis; Gall Stone
MeSH Terms: conditions — Liver Cirrhosis; Gallstones

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genetic Analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cirrhosis with GSD: Cirrhosis with GSD
- No cirrhosis with no GSD: No cirrhosis with no GSD
- Cirrhosis with no GSD: Cirrhosis with no GSD
- GSD with no cirrhosis: GSD with no cirrhosis
- Cirrhosis with history of cholecystectomy for GSD: Cirrhosis with history of cholecystectomy for GSD

SUMMARY:
Gall stone disease is more common in patients with cirrhosis. This association has been well established in different studies. Among the various factors which predispose a patient with gall stone disease to have associated liver cirrhosis, genetics also plays an important role.

This study aims to do a genetic panel-based analysis of genes which are involved in cholestasis to find any association between liver cirrhosis and gall stone disease.

Patients with history of gall stone or history of cholecystectomy done for gall stone disease will be evaluated for the presence of liver cirrhosis by fibroscan and ultrasonography. Those patients with cirrhosis and without cirrhosis will undergo a panel based genetic test for the common cholestasis genes and multivariate analysis will be done for variants associated with lithogenesis and cirrhosis.

DETAILED DESCRIPTION:
Study population:

* Patients > 18 years of age.
* Who have either gall stone disease or cirrhosis. Study design: All consecutive in-patients and out-patients requiring liver biopsy for evaluation of diffuse parenchymal liver disease will be evaluated for inclusion.

Study period: 1 year. Intervention: Blood sample from included patients will be subject to panel based NGS.

Monitoring and assessment: History of all patients including family history will be taken. Screening for cirrhosis will be done by fibroscan or ultrasound scanning. Gall stone diagnosis is made by USG. History about patients' parents, siblings, spouse, children will be taken with respect to gall stone and cirrhosis. NGS of cholecystitis will be send for the subject and the results will be collected as the fastQ file for analysis.

Statistical Analysis: MVA will be done to identify gene variants independently associated with lithogenesis and cirrhosis, along with demographic and environmental risk factors for these conditions. * From this data, overlapping risk-variants in common associated genes will be identified. A risk estimate (OR with 95% CI) will be calculated for each of the above identified genetic risk variant for the phenotype of cirrhosis with GS.

Adverse effects:

There are no adverse outcomes with respect to this study. Stopping rule of study: There are no stopping rules for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years of age.
2. Who has a GSD diagnosed by USG or have history of cholecystectomy for gall stone disease.
3. Who is a diagnosed case of cirrhosis by Fibroscan or USG (Cirrhosis including alcohol related cirrhosis, Hepatitis B, Hepatitis C, Wilsons disease, Hemochromatosis are excluded.

Exclusion Criteria:

1. Patients who have haemolytic anaemia
2. Patients who do not consent for genetic study
3. Patients who has a diagnosed cause for liver disease, including alcohol related cirrhosis, Hepatitis B, Hepatitis C, Wilsons disease, Hemochromatosis.
4. Inability to provide informed consent.
5. Cannot understand Hindi or English should be excluded since they will not be able to reply objectively to questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients > 18 years of age.
  * Who have either gall stone disease or cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic risk-variants associated with both GS and modulation of liver cirrhosis in patients with cirrhosis. | Day 0

SECONDARY OUTCOMES:
Identification of genetic polymorphisms in bile-acid metabolism and enterohepatic circulation, associated with increased GS risk in patients with cirrhosis. | Day 0
Identification of genetic polymorphisms in cholesterol metabolism pathway, associated with increased GS risk in patients with cirrhosis. | Day 0
To study the association of UGT1A1 polymorphisms affecting bilirubin conjugation, with risk of GS in patients with cirrhosis. | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided